CLINICAL TRIAL: NCT03887871
Title: An Open-label, Randomized, Fed, Single Dose, Crossover Study to Evaluate the Bioequivalence of Chong Kun Dang Pharmaceutical "Chong Kun Dang Tamsulosin HCl Tablet" and Astellas Phama Korea Inc. "Harnal-D" in Healthy Volunteers
Brief Title: Study to Evaluate the Bioequivalence of Astellas Phama Korea Inc. "Harnal-D" in Healthy Volunteers After Meal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BE117721820/DDS18-030BE
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference/Test (Experimental): 1. Period 1: Harnal-D Tab. 1T
  2. Period 2: Chong Kun Dang Tamsulosin HCl Tab. 1T
  Interventions: Drug: Harnal-D Tab.; Drug: Chong Kun Dang Tamsulosin HCl Tab.
- Test/Reference (Experimental): 1. Period 1: Chong Kun Dang Tamsulosin HCl Tab. 1T
  2. Period 2: Harnal-D Tab. 1T
  Interventions: Drug: Harnal-D Tab.; Drug: Chong Kun Dang Tamsulosin HCl Tab.

INTERVENTIONS:
Drug: Harnal-D Tab. — Harnal-D Tab. 1T single oral administration after meal
Drug: Chong Kun Dang Tamsulosin HCl Tab. — Chong Kun Dang Tamsulosin HCl Tab. 1T single oral administration after meal

SUMMARY:
This study is an open-label, randomized, fed, single dose, crossover study to evaluate the bioequivalence of Chong Kun Dang Pharmaceutical "Chong Kun Dang Tamsulosin HCl Tablet" and Astellas Phama Korea Inc. "Harnal-D" in healthy volunteers

DETAILED DESCRIPTION:
To healthy subjects of thirty (30), following treatments are administered dosing in each period and wash-out period is a minimum of 1 week.

Reference drug: Harnal-D Tab. / Test drug: Chong Kun Dang Tamsulosin HCl Tab. Pharmacokinetic blood samples are collected up to 48hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject older than 19 years men at the screening
2. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination(if necessary, EEG, ECG, chest X-ray, endoscope or upper gastrointestinal radiography)
3. Individuals who were deemed to be appropriate as study subjects in accordance with the screening results (laboratory tests, ECG etc.)
4. Individuals who had 18 kg/m2 ≤ Body Mass Index(BMI) ≤ 30kg/m2

   * BMI = Weight(kg)/ Height(m)2
5. Individuals who had agreed to participate in the study
6. Individuals without mental illness history within five year prior to the screening
7. Individuals without a medical history of gastrointestinal operations that may affect drug absorption
8. Individuals who do not agree to the approved methods of double contraception and using spermicide for up to 7 days after investigational product(s) administration

Exclusion Criteria:

1. Individuals who had enrolled to barbiturate's drugs by induction and inhibition of drug-metabolizing enzymes of drugs within the 1 month
2. Individuals who had excessive drinking within the 1 month

   *Men: 21 glasses/week exceeded(1 glass: distilled spirits 45 mL, wine 150 mL, beer 360 mL)
3. Individuals who had taken any medication within 10 days prior to the first day of dosing
4. Individuals who were deemed to be inappropriate to participate in the study by the investigator
5. Individuals who had participated of other clinical study or bioequivalence study within the 3 months prior to the first day of dosing
6. Individuals who donated whole blood within the 2 months, or blood components within 1 weeks prior to the first dose of the investigational product(s)
7. Individuals with hypersensitivity (include Vascular edema) to ingredients used in the investigational product(s)
8. Individuals with hereditary diseases of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption etc.
9. Individuals with orthostatic hypotension
10. Individuals with severe hepatopathy
11. Individuals who had taken alpha-1 blocker
12. Individuals who had history of micturition syncope
13. Individuals with nephropathy
14. Elderly person
15. Individuals who had taken PDE5(phosphodiesterase-5) inhibitor
16. Individuals who had taken CYP3A4 inhibitor
17. Individuals who had taken antihypertensive drug(s)

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
AUCt of Chong Kun Dang Tamsulosin HCl Tablet and Harnal-D | Pre-dose (0 hour), post-dose 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 hours
  Area under the Chong Kun Dang Tamsulosin HCl Tablet / Harnal-D concentration in blood-time curve from zero to final
Cmax of Chong Kun Dang Tamsulosin HCl Tablet and Harnal-D | Pre-dose (0 hour), post-dose 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 48 hours
  The maximum Chong Kun Dang Tamsulosin HCl Tablet / Harnal-D concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jung Cha, Principal Investigator — Bestian Hospital
Locations (1):
- Bestian Hospital, Osŏng, South Korea

IPD SHARING:
Plan to Share IPD: No